CLINICAL TRIAL: NCT00004297
Title: Phase III Randomized Study of Diazepam Vs Lorazepam Vs Placebo for Prehospital Treatment of Status Epilepticus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: University of California, San Francisco (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11733; UCSF-69020732504A
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Status Epilepticus
Keywords: epilepsy; neurologic and psychiatric disorders; rare disease; seizures; status epilepticus
MeSH Terms: conditions — Status Epilepticus; Epilepsy; Neurologic Manifestations; Mental Disorders; Rare Diseases; Seizures | interventions — Diazepam; Lorazepam

INTERVENTIONS:
Drug: diazepam
Drug: lorazepam

SUMMARY:
OBJECTIVES: I. Compare the efficacy, onset of clinical anticonvulsant activity, and complications of diazepam and lorazepam given intravenously as prehospital therapy to patients in status epilepticus.

II. Determine the effect of prehospital therapy on the incidence of status epilepticus at the subsequent emergency department admission.

III. Establish whether prehospital therapy alters hospital management of these patients and ultimately affects patient outcome.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, multicenter study. Patients are stratified by center.

Patients en route to the hospital in a San Francisco Department of Health Paramedic Division ambulance are randomly assigned to 1 of 3 treatment groups. Informed consent is waived due to impaired consciousness.

Patients receive intravenous diazepam, lorazepam, or placebo during transport. The patient is re-treated if the seizure is sustained after the first dose or recurs after the first dose without the patient regaining consciousness.

Upon arrival at the hospital, all patients receive the standard status epilepticus treatment in use at that site.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Status epilepticus with at least 5 minutes of sustained seizure activity with a depressed level of consciousness, or 2 or more discrete seizures without recovery or consciousness between seizures Verified by bystander or observed by paramedic from San Francisco Department of Health --Prior/Concurrent Therapy-- No chronic benzodiazepines for seizure disorder --Patient Characteristics-- Cardiovascular: Systolic blood pressure at least 100 mm Hg No second- or third- degree atrioventricular block No sustained ectopic tachyrhythmia Pulse rate between 60 and 150 No severe myocardial insufficiency No hypovolemic, cardiogenic, or obstructive shock Pulmonary: No history of asthma No history of chronic obstructive airway disease No history of limited pulmonary reserve Other: No allergy or prior sensitivity to benzodiazepines No distributive shock (e.g., septic, neurogenic, or anaphylactic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210
Dates: Start 1995-11; Study Completion 1999-02

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lowenstein, Study Chair — University of California, San Francisco